CLINICAL TRIAL: NCT00082485
Title: Multi-Center Trial of Baclofen for the Treatment of Cocaine Dependence
Brief Title: Baclofen for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Liza Gorgon, National Institute on Drug Abuse
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-CSP-1021-1; NCT00431938 (obsolete NCT alias)
Record Dates: First submitted 2004-05-11; First posted 2004-05-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-08

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Baclofen
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Baclofen — Dose escalation 10-60mg (week 1) 60 mg (weeks 2-7) Dose taper (week 8)
  Arms: 1
Other: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy and safety of baclofen for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
Double-blind, placebo-controlled, parallel design trial of baclofen for the treatment of cocaine dependence

ELIGIBILITY:
Inclusion Criteria:

* Subject must have DSM-IV diagnosis of cocaine dependence.
* Subject must be seeking treatment for cocaine dependence.
* Be be able to verbalize understanding of consent form, provide written consent and verbalize willingness to complete study procedures.

Exclusion Criteria:

* Please contact site for more information.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-06; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Effects of medication on cocaine craving

CONTACTS AND LOCATIONS:
Overall Officials: Liza Gorgon, M.A., Principal Investigator — VA Maryland Health Care System
Locations (8):
- United States (8):
  - San Francisco General Hosptial, San Francisco, California
  - Torrance Site, Torrance, California
  - Denver VA Medical Center, Denver, Colorado
  - VA Maryland Healthcare System, Baltimore, Maryland
  - U of Penn School of Medicine, Philadelphia, Pennsylvania
  - South TX VA Health Care System, San Antonio, Texas
  - Salt Lake City VA Medical Center, Salt Lake City, Utah
  - Institute of Resch & Educ Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Result] Kahn R, Biswas K, Childress AR, Shoptaw S, Fudala PJ, Gorgon L, Montoya I, Collins J, McSherry F, Li SH, Chiang N, Alathari H, Watson D, Liberto J, Beresford T, Stock C, Wallace C, Gruber V, Elkashef A. Multi-center trial of baclofen for abstinence initiation in severe cocaine-dependent individuals. Drug Alcohol Depend. 2009 Jul 1;103(1-2):59-64. doi: 10.1016/j.drugalcdep.2009.03.011. Epub 2009 May 2. PMID 19414226